CLINICAL TRIAL: NCT02552927
Title: Effect of Chest Shielding on the Incidence of Patent Ductus Arteriosus in Premature Infants Undergoing Phototherapy
Brief Title: Chest Shielding in Premature Infants During Phototherapy
Acronym: SLIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 55472; 911 (Other: Urochester)
Record Dates: First submitted 2015-08-17; First posted 2015-09-17 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Patent Ductus Arteriosus in Premature Infants
Keywords: PDA; Jaundice; Phototherapy
MeSH Terms: conditions — Jaundice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CALF (Experimental): Chest shield with aluminum foil
  Interventions: Device: Chest shield with aluminum foil (CALF)
- SHIELD (Sham Comparator): Chest shield without aluminum foil
  Interventions: Device: SHIELD

INTERVENTIONS:
Device: Chest shield with aluminum foil (CALF)
  Arms: CALF
Device: SHIELD
  Arms: SHIELD

SUMMARY:
This is a feasibility study where Infants will be randomized to either chest shielding with aluminum foil or chest shielding without aluminum foil while undergoing phototherapy for premature infants. The primary outcome is patent ductus arteriosus.

ELIGIBILITY:
Inclusion Criteria:

* less or equal to 29 weeks or 1000g at birth
* Admitted to the NICU (Neonatal intensive care unit) within 24 hours after birth
* English speaking parents

Exclusion Criteria:

* Congenital abnormalities
* Chromosomal disorders
* Cyanotic heart defects
* Nitric oxide
* Prophylactic phototherapy
* Unlikely to survive beyond 72 hours according to the attending neonatologist
* Do not require phototherapy

Ages: 23 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic Patent ductus arteriosus | During first 2 weeks

SECONDARY OUTCOMES:
Urinary Nitric oxide level | During first 2 weeks

OTHER OUTCOMES:
Incidence of Chronic lung disease | at 36 weeks post-menstrual age
Incidence of Retinopathy of Prematurity | up to 44 weeks post-menstrual age
Peak level of total serum bilirubin | First 2 weeks
Duration of Phototherapy | First 2 weeks
Incidence of intraventricular hemorrhage | First 2 weeks
Incidence of surgical ligation for patent ductus arteriosus | First 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Javed Mannan, MD, MPH, Study Director — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Mannan J, Amin SB. Effect of chest shielding during phototherapy for hyperbilirubinemia on symptomatic patent ductus arteriosus - a double-blind randomized placebo-controlled trial. Pediatr Res. 2024 Dec;96(7):1771-1776. doi: 10.1038/s41390-024-03310-4. Epub 2024 Jun 22. PMID 38909157